CLINICAL TRIAL: NCT02034279
Title: Albumin Administration in the Prevention of Hepatorenal Syndrome and Death in Patients With Cirrhosis, Bacterial Infections Other Than Spontaneous Bacterial Peritonitis and High Risk of Hospital Mortality
Brief Title: The INFECIR-2 Albumin Prevention Study
Acronym: INFECIR2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment rate and expiration of the study drug
Sponsor: EASL - CLIF Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INFECIR 2; 2013-002416-27 (EudraCT Number)
Record Dates: First submitted 2014-01-07; First posted 2014-01-13 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Advanced Chronic Liver Disease; Urinary Infection; Pneumonia; Cholangitis; Other Bacterial Diseases
Keywords: cirrhosis
MeSH Terms: conditions — Urinary Tract Infections; Pneumonia; Cholangitis; Fibrosis | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous infusion of albumin (Experimental): Treatment arm will receive intravenous albumin on days 1 and 3 plus antibiotics
  Interventions: Drug: Albumin
- No albumin (No Intervention): Only antibiotics

INTERVENTIONS:
Drug: Albumin — Intravenous infusion of 20% albumin
  Other Names: Albutein 20 by Grifols
  Arms: Intravenous infusion of albumin

SUMMARY:
The aim of this study is to evaluate whether albumin administration improves short-term survival in patients with advanced cirrhosis and bacterial infections other than Spontaneous Bacterial Peritonitis (SBP).

DETAILED DESCRIPTION:
The aim of this study is to evaluate if IV albumin administration improves short-term survival in patients with advanced cirrhosis (serum creatinine ≥ 1.2 mg/dl, serum sodium ≤ 130 mEq/l -milliequivalents per liter- and/or serum bilirubin ≥4 mg/dl) and bacterial infections other than spontaneous bacterial peritonitis (urinary infection, pneumonia, spontaneous or secondary bacteremia, skin/soft tissue infection, acute cholangitis or suspected bacterial infection).

Primary goals of the study:

• Effect of albumin administration on hospital survival

Secondary goals of the study:

* Effect of albumin administration on 28-day and 90-day survival.
* Effect of albumin administration on the incidence of renal dysfunction, AKI, type-1 and 2 Hepatorenal Syndrome (HRS) during hospitalization.
* Effect of albumin on circulatory function estimated by changes in plasma levels of renin and noradrenaline and in serum levels of lactate among infection diagnosis, day 3 and infection resolution.
* Effect of albumin on serum levels of interleukin-6 (IL-6), tumor necrosis factor alpha (TNF-alpha) and nitric oxide (NOX) and on plasma levels of von Willebrand factor (vWF:Ag) at diagnosis and resolution of infection.
* Effect of albumin on blood leukocyte count and serum C-reactive protein levels (CRP) during infection.
* Effect of albumin on the development of other individual organ failures (renal, liver, cerebral, circulatory, coagulation and respiratory), acute-on-chronic liver failure (ACLF type 1, 2 and 3 according to the Canonic Study), CLIF-SOFA score, CLIF-Consortium score, Child-Pugh score and MELD score during hospitalization.
* Evaluation of predictive factors of HRS and ACLF development in non-SBP infections.
* Samples (blood, plasma, serum and urine) will be obtained and stored for genomic, proteomic and standard biochemical investigations in future ancillary studies related to the aim of the study.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients with age ≥18 years
* Diagnosis of urinary infection, pneumonia, spontaneous or secondary bacteremia, skin/soft tissue infection, acute cholangitis or suspected bacterial infection at hospital admission or during hospitalization
* Patients with uncomplicated urinary infections or suspected bacterial infection will require the presence of signs of systemic inflammation: at least 1 diagnostic criterion of systemic inflammatory response syndrome (SIRS) and serum CRP levels ≥1 mg/dl (10 mg/L). This criterion will not be required for the rest of infections
* Analytical data of renal and/or liver dysfunction (serum creatinine ≥ 1.2 mg/dl, serum sodium ≤ 130 mEq/l, serum bilirubin ≥4 mg/dl). Patients with pneumonia or documented bacteremia (positive blood cultures) will require the presence of at least 1 of these analytical criteria to be included in the study. Patients with urinary infection, skin/soft tissue infection, acute cholangitis or suspected bacterial infection will require 2 or more criteria for inclusion

Exclusion Criteria:

* > 72h after infection diagnosis
* Pregnancy
* Acute or subacute liver failure without underlying cirrhosis
* Septic shock
* Severe acute respiratory distress syndrome (Pa02/Fi02 ≤ 100)
* Active or recent variceal bleeding unless controlled for > 48h
* Ongoing type-1 HRS (past IAC criterion: serum creatinine ≥ 2.5 mg/dl)
* Type-3 ACLF (defined according to the Canonic Study criteria)
* Hemodialysis or other renal replacement therapy
* Evidence of current malignancy (except for hepatocellular carcinoma within Milan criteria or non-melanocytic skin cancer)
* Moderate or severe chronic heart (NYHA class II, III or IV) or pulmonary disease (GOLD IV)
* Severe psychiatric disorders
* Previous liver transplantation
* HIV infection (except for patients under antiretroviral therapy with undetectable viral load, CD4>200/mm3 and no history of opportunistic infections diagnostic of AIDS)
* Contraindications to albumin (allergy, signs of pulmonary edema)
* Albumin administration (≥ 80g) in the last 2 days
* Spontaneous bacterial peritonitis coinfection
* Use of any investigational drug within 90 days prior to randomization
* Refusal to participate
* Patients who cannot provide prior informed consent and when there is documented evidence that the patient has no legal surrogate decision maker and it appears unlikely that the patient will regain consciousness or sufficient ability to provide delayed informed consent
* Physician and team not committed to intensive care if needed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
survival | hospitalization
  Hospital survival will be the primary outcome

SECONDARY OUTCOMES:
survival | 28-d and 90-day survival
  Percentage of subjects within each arm that survived at these time points
Renal dysfunction | hospitalization (expected average 2 weeks)
  number of participants
circulatory dysfunction | day 3 and day of infection resolution
  plasma concentration of hormones
Inflammation and endothelial function | day of infection resolution
  Plasma concentration of cytokines
subsequent organ failure | hospitalization (expected average 2 weeks)
  number of organ failures

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Gustot, Principal Investigator — Erasme University Hospital, Brussels, Belgium; Frederick Nevens, Principal Investigator — University Hospitals KU, Leuven, Belgium; Faouzi Saliba, Principal Investigator — Hôpital Paul Brousse, Villejuif, France; François Durand, Principal Investigator — Hôpital Beaujon, Clichy, France; Matthias Dollinger, Principal Investigator — University of Ulm, Heidelberg and Tübingen, Germany; Stefan Zeuzem, Principal Investigator — University Hospital of Frankfurt, Germany; Alexander Gerbes, Principal Investigator — University Hospital of Munich, Germany; Jonel Trebicka, Principal Investigator — University Hospital of Bonn, Germany; Henning Gronbaeck, Principal Investigator — Aarhus University Hospital; Fin Stolze Larsen, Principal Investigator — Rigshospitalet, University of Copenhagen; John Willy Haukeland, Principal Investigator — Oslo University Hospital; Andrea de Gottardi, Principal Investigator — Bern University Hospital, Switzerland; Aide McCormick, Principal Investigator — University College of Dublin, Ireland; Rajiv Jalan, Principal Investigator — University College, London; Marco Domenicali, Principal Investigator — Santa Orsola-Malpighi Hospital, Bologna, Italy; Paolo Angeli, Principal Investigator — University of Padova, Italy; Carlo Alessandria, Principal Investigator — San Giovanni Battista Hospital, University of Turin, Italy; Francesco Salerno, Principal Investigator — Policlinico IRCCS San Donato, University of Milan, Italy; Agustin Albillos, Principal Investigator — Hospital Ramon y Cajal, Madrid, Spain; Victor Vargas, Principal Investigator — Hospital Vall d'Hebron, Barcelona, Spain; Javier Fernandez, Principal Investigator — Hospital Clinic, Barcelona, Spain; German Soriano, Principal Investigator — Hospital Santa Creu i Sant Pau, Barcelona, Spain; Rafael Bañares, Principal Investigator — Hospital Gregorio Marañon, Madrid, Spain; Jose Luis Montero, Principal Investigator — Hospital Reina Sofia, Cordoba, Spain; Manuela Merli, Principal Investigator — Sapienza University of Rome, Italy; Minneke Coenraad, Principal Investigator — Leiden University Medical Center; Rudolf Stauber, Principal Investigator — Medical University of Graz; Wolfgang Vogel, Principal Investigator — Medical Hospital Innsbrück
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet

REFERENCES:
- [Background] Guevara M, Terra C, Nazar A, Sola E, Fernandez J, Pavesi M, Arroyo V, Gines P. Albumin for bacterial infections other than spontaneous bacterial peritonitis in cirrhosis. A randomized, controlled study. J Hepatol. 2012 Oct;57(4):759-65. doi: 10.1016/j.jhep.2012.06.013. Epub 2012 Jun 23. PMID 22732511
- [Background] Thevenot T, Bureau C, Oberti F, Anty R, Louvet A, Plessier A, Rudler M, Heurgue-Berlot A, Rosa I, Talbodec N, Dao T, Ozenne V, Carbonell N, Causse X, Goria O, Minello A, De Ledinghen V, Amathieu R, Barraud H, Nguyen-Khac E, Becker C, Paupard T, Botta-Fridlung D, Abdelli N, Guillemot F, Monnet E, Di Martino V. Effect of albumin in cirrhotic patients with infection other than spontaneous bacterial peritonitis. A randomized trial. J Hepatol. 2015 Apr;62(4):822-30. doi: 10.1016/j.jhep.2014.11.017. Epub 2014 Nov 21. PMID 25463545
- [Derived] Fernandez J, Angeli P, Trebicka J, Merli M, Gustot T, Alessandria C, Aagaard NK, de Gottardi A, Welzel TM, Gerbes A, Soriano G, Vargas V, Albillos A, Salerno F, Durand F, Banares R, Stauber R, Prado V, Arteaga M, Hernandez-Tejero M, Aziz F, Morando F, Jansen C, Lattanzi B, Moreno C, Campion D, Gronbaek H, Garcia R, Sanchez C, Garcia E, Amoros A, Pavesi M, Claria J, Moreau R, Arroyo V. Efficacy of Albumin Treatment for Patients with Cirrhosis and Infections Unrelated to Spontaneous Bacterial Peritonitis. Clin Gastroenterol Hepatol. 2020 Apr;18(4):963-973.e14. doi: 10.1016/j.cgh.2019.07.055. Epub 2019 Aug 5. PMID 31394283
- See also: Web page of the INFECIR-2 RCT — http://www.clifresearch.com/infecir2/Home.aspx